CLINICAL TRIAL: NCT03510533
Title: Validation of the Concept of the Autoantibodies Directed Against the Neuropeptides Involved in Food Intake Regulation on the Incidental Cases of Eating Disorders
Acronym: EDILS-AutoAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016/0107/HP; 2017-A00875-48 (Other: Agence Nationale de Sécurité du médicament et des produits de Santé)
Record Dates: First submitted 2018-04-04; First posted 2018-04-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Eating Disorder
Keywords: autoantibodies (autoAc) circulating; neuropeptides (Ghrelin, l'α-MSH); potential digestive origin
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Ghrelin; alpha-MSH; Appetite Regulation; Endopeptidase Clp

STUDY DESIGN:
Intervention Model Description: Eating disorders compared to healthy volonteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eating disorders patients (Experimental): first clinical visit in nutrition department of CHU de Rouen for eating disorders (anorexia nervosa, hyperphagia or bulimia) according to the classification DSM-V
  Interventions: Other: Evaluation of the rates of the autoantibodies directed against the neuropeptides (ghrelin and alpha-MSH) controlling involved in food intake regulation
- healthy volunteers (Other): Volunteers with negative SCOFF test (No active or history of eating disorders)
  Interventions: Other: Evaluation of the rates of the autoantibodies directed against the neuropeptides (ghrelin and alpha-MSH) controlling involved in food intake regulation

INTERVENTIONS:
Other: Evaluation of the rates of the autoantibodies directed against the neuropeptides (ghrelin and alpha-MSH) controlling involved in food intake regulation — blood samples (12ml) and stool samples (30g) collections
  Other Names: Evaluation of the rate of the autoantibodies directed against bacterial peptide, ClpB; Factors associated with eating disorders

SUMMARY:
This study should lead to the validation of the concept of the autoAc directed against the neuropeptides involved in food intake regulation.

DETAILED DESCRIPTION:
Eating disorders are a public health issue. It has been recently reported the importance of immune system modifications in eating disorders physiopathology, involving autoantibodies directed against neuropeptides regulating food intake. A recent study of laboratory INSERM 1073 showed the existence of an intestinal bacterial protein exhibiting structural similarities with α-MSH: ClpB. The autoAc directed against the latter also react with α-MSH because of these similarity of structures, thus leading to a potential digestive origin of these autoAc. To consolidate this new etiopathogenic assumption, a large clinical study is necessary with analysis of patients autoAc profiles. a monocentric study with inclusion of 240 patients over 2 years and 80 healthy volunteers is proposed.

This study should lead to the validation of the concept of the autoAc directed against the neuropeptides involved in food intake regulation. Nutritional modulations (probiotic, amino-acid…) could constitute an interesting therapeutic perspective in the future.

ELIGIBILITY:
Inclusion Criteria:

Patients with eating disorders

1. 18 Years and older
2. first clinical visit in nutrition department of CHU de Rouen for eating disorders
3. anorexia nervosa, hyperphagia or bulimia according to the classification DSM-V
4. social security Affiliation
5. Patient who signed the MEC approved informed consent

Volunteers

1. 18 Years to 60 Years
2. body mass index ≥ 18,5 kg/m2 and ≤ 24,9 kg/m2
3. negative SCOFF test
4. No active and history of eating disorders
5. social security Affiliation
6. volunteer who signed the MEC approved informed consent

Exclusion criteria:

Patients with eating disorders

1. No anorexia nervosa, hyperphagia or bulimia according to the classification DSM-V
2. Adults under legal protection or under safeguard of justice or administrative decision
3. Pregnancy

Volunteers

1. Active or history of eating disorder
2. Adults under legal protection or under safeguard of justice or administrative decision
3. Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 211 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of the rates of the autoantibodies directed against the neuropeptides (ghrelin and alpha-MSH) involved in food intake regulation among patients with eating disorders | 1 week
  blood samples collections

SECONDARY OUTCOMES:
Scale for determination factors associated with eating disorders | 1 week
  A global scale will evaluate :
  * socio demographic factors
  * somatic and psychiatric comorbidities
  * addictions
  * personal and family antecedents
  * major events
statute in autoantibody and behavioral characteristics of the eating disorder | 1 week
  quality of life and the psychological state of the patients tests
Evaluation of the rate of the autoantibodies directed against bacterial peptide, ClpB among patients presenting with eating disorders | 1 week
  stoll samples collections

CONTACTS AND LOCATIONS:
Overall Officials: Najate EL MACHKOURI ACHAMRAH, MD, PhD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Centre d'Investigation Clinique, Rouen, France